CLINICAL TRIAL: NCT03191903
Title: Randomized, Double-Blind, Active Comparator Controlled, Multi-Center Study of a Single Injection Cross-Linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (Cingal™) to Provide Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Study of Cingal™ for the Relief of Knee Osteoarthritis Compared to Triamcinolone Hexacetonide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cingal 16-02
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Intra-articular Injection; Hyaluronic Acid; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — 3,6,9,16,19,22-hexaaza-6,19-bis(2-hydroxyethyl)tricyclo(22,2,2,2(11,14))triaconta-1,11,13,24,27,29-hexaene; triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in a 4:4:1 ratio into the Cingal, Monovisc (hyaluronic acid) or TH (triamcinolone hexacetonide) arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study subjects and the Outcomes Assessor are blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Cingal (Experimental): Cingal is a combination product consisting of 88 milligrams of cross-linked HA (hyaluronic acid) with 18 milligrams of TH (triamcinolone hexacetonide) in a 4 milliliter (mL) intra-articular injection.
  Interventions: Combination Product: Cingal
- Monovisc (Active Comparator): Monovisc is a device that consists of 88 milligrams of cross-linked HA (hyaluronic acid) in a 4 milliliter (mL) intra-articular injection.
  Interventions: Device: Monovisc
- Triamcinolone Hexacetonide (TH) (Active Comparator): Triamcinolone hexacetonide (TH) is a corticosteroid supplied in a 20 milligram per 1 milliliter (20 mg/mL) intra-articular injection.
  Interventions: Drug: Triamcinolone Hexacetonide

INTERVENTIONS:
Combination Product: Cingal — Hyaluronic Acid with Triamcinolone Hexacetonide
  Other Names: HA + TH
  Arms: Cingal
Device: Monovisc — Hyaluronic acid
  Other Names: HA
  Arms: Monovisc
Drug: Triamcinolone Hexacetonide — Triamcinolone Hexacetonide
  Other Names: TH
  Arms: Triamcinolone Hexacetonide (TH)

SUMMARY:
This is a multi-center, randomized, double-blind, parallel group, active comparator controlled trial to evaluate the efficacy and safety of a single injection of Cingal for the relief of joint pain in subjects with OA of the knee.

DETAILED DESCRIPTION:
Cingal 16-02 is a multi-center, randomized, double-blind, active comparator controlled study designed to evaluate the relative contributions of the individual constituents (Hyaluronic Acid and Triamcinolone Hexacetonide) in the Cingal combination product to pain relief as measured by the change in WOMAC Pain from baseline through 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

Screening Inclusion Criteria

1. Subject is 40-75 years old, with a Body Mass Index (BMI) ≤ 40 kg/m2.
2. Subject has Kellgren-Lawrence (K-L) severity grade I, II or III in the index knee as determined by X-ray. Contralateral knee: K-L severity grade 0, I or II.
3. Subject has had at least two signs and at least two symptoms of OA disease (based on the European League Against Rheumatism (EULAR) recommendations for diagnosing knee OA) in the index knee for at least 6 months despite conservative treatment (weight reduction, physical therapy, pain medications, etc.). The EULAR signs and symptoms are as follows:

   * Signs: crepitus, restricted movement and bony enlargement
   * Symptoms: persistent knee pain, limited morning stiffness and reduced function
4. Subject must be willing to abstain from other IA treatments of the knee for the duration of the study.
5. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
6. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty eight hours prior to the Baseline Visit and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol.
7. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
8. Subject is able to understand and comply with the requirements of the study and voluntarily provides consent.

Screening Exclusion Criteria:

1. Subject received an IA injection of Hyaluronic Acid (HA) and/or steroid in either knee within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either knee during the course of this study.
2. Subject had an arthroscopy of either knee within 3 months of signing the ICF.
3. Subject had an open surgical procedure of either knee or hip or any surgery of the spine within 12 months of signing ICF. Subject plans to have knee, hip or spine surgery within the study period.
4. Subject has intra-articular trauma to the index knee. Subject has concurrent multi-system or multi-limb trauma.
5. Subject has evidence or medical history of the following diseases in the index knee: septic arthritis; inflammatory joint disease; history of Reiter's syndrome; gout; chondrocalcinosis associated with recurrent episodes of acute synovitis of the knee consistent with pseudogout; osteochondritis dissecans, Paget disease of the bone; ochronosis; acromegaly; hemochromatosis; primary osteochondromatosis; known history of Wilson disease; heritable disorders or collagen gene mutations.
6. Subject has a history of cartilage repair surgery in the index knee within 3 years of signing the ICF.
7. Subject has a history of ACL repair, reconstruction or injury in the index knee within 3 years of signing the ICF.
8. Subject has X-ray findings of acute fractures, severe bone loss, avascular necrosis, severe bone or joint deformity in the index knee.
9. Subject has significant varus or valgus deformity greater than 10 degrees in either knee.
10. Subject has a clinically apparent tense effusion of the index knee.
11. Subject has knee instability in either knee per the Investigator's assessment.
12. Subject requires consistent use of an assistive device (e.g. wheelchair, walker, etc.) Occasional use of a cane is acceptable.
13. Subject has medical condition(s) which could affect study assessments or may adversely affect the safety and/or success of the study treatment. This includes but is not limited to the following: a. Peripheral neuropathy severe enough to interfere with evaluation of the subject, b. Vascular insufficiency severe enough to interfere with evaluation of the subject, c. Active fibromyalgia, d. Hemiparesis involving either lower extremity, e. Immunocompromised or immunosuppressive disorder or receiving medications to treat immunosuppressive disorders, f. Systemic bleeding disorder(s), g. Current malignancy or treatment within the last 5 years, except for non-melanoma skin cancer, h. Significant psychiatric disorder, i. Active drug and/or alcohol abuse within the past year, j. Uncontrolled diabetes with a screening HbA1c of >7%.
14. Subject is taking medications at the time the subjects signs the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
15. Subject is receiving treatment using electromagnetic stimulation and/or low intensity ultrasound in the index knee at the time of signing the ICF, within 3 months of signing the ICF or plans to receive treatment any time during the study period.
16. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index knee only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index knee is allowed.
17. Subject has a pre-treatment contraindication to IA injections or aspiration of the index knee, including cutaneous infection in the injection site area, active IA infection (as suggested by moderate or marked effusion), knee deformity or condition which, in the opinion of the Investigator could jeopardize the sterility or delivery of the IA injection.
18. Subjects with a history of hypersensitivity to any of the ingredients in the hyaluronan or previous hypersensitivity to the administration of corticosteroids or an inability to tolerate acetaminophen/paracetamol.
19. Subject has any contraindication to the receipt of a corticosteroid.
20. Subject is receiving or in litigation for worker's compensation.
21. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
22. Subject was involved in any other research study involving an investigational product, or a new application of an approved product, within 60 days of signing the ICF.

Baseline Inclusion Criteria:

1. Subject has a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain-sub-score ≥ 40 mm and ≤ 90 mm in the affected knee and ≤ 30 mm in the contralateral knee on a 100 mm Visual Analog Scale (VAS) scale.

Baseline Exclusion Criteria:

1. Subject has a decrease of ≥ 20 mm in the WOMAC pain-sub-score (average of 5 pain scales) from Screening to Baseline in the index knee on a 100 mm Visual Analog Scale (VAS) scale.
2. Subject has a synovial fluid aspirate volume > 20 mL in the index knee.
3. Subject has a contraindication to continue with the study treatment injection based on the visual appearance of the synovial fluid aspirate unless the fluid is examined microscopically prior to injection with no clinically significant findings (e.g. bacteria, crystals or blood).
4. Subject has range of motion of less than 100° flexion in either knee.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, Principal Investigator — Uzsoki Hospital, Department of Traumatology
Locations (19):
- Hungary (8):
  - Health Center of Downtown-Lipotvaros, Orthopedic Outpatient Clinic (Belvárosi-Lipótvárosi Egészségügyi Szolgálat Ortopeadia), Budapest
  - Magyar Honvedseg, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Baleseti Központ, Budapest
  - DE KK Ortopediai Klinika, Debrecen
  - Jutrix Medical Llc, Kecskemét
  - Medidea Bt., Kiskunfélegyháza
  - Kastelypark Klinka, Tata
- Poland (11):
  - Zdrowie Osteo-Medic, Bialystok
  - Szpital Świętego Łukasza S.A., Bielsko-Biala
  - NZOZ Medi SPATZ, Gliwice
  - ARTIMED Niepubliczny Zakład Opieki Zdrowotnej, Kielce
  - Centrum Medyczne 4M Plus, Krakow
  - Medical University of Lodz, Lodz
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - NOVAMED Jackowiak Krajewski Spółka Jawna, Torun
  - Centrum Medyczne Amed Warszawa Targówek, Warsaw
  - ETG Network, Warsaw, Warsaw
  - ETG Network, Warsaw

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at trial sites into the Cingal 16-02 study in May 2017 through September 2017.
Pre-assignment Details: One participant met the screening eligibility criteria but failed the baseline screening criteria due to aspirate criteria. This subject was not treated.
Period: Overall Study
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Started (Safety Population) | 251 | 251 | 74
Intent to Treat Population | 251 | 251 | 74
Completed | 244 | 246 | 70
Not Completed | 7 | 5 | 4
Not completed — Withdrawal by Subject | 6 | 5 | 4
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety and Intent to Treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH) | Total
Number analyzed (Participants) | 251 | 251 | 74 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (8.7) | 57.7 (8.9) | 59.0 (8.5) | 58.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 163 | 52 | 394
  Male | 72 | 88 | 22 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 251 | 251 | 74 | 576
Baseline WOMAC Pain in Index Knee [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score is a validated scale from 0 to 100 mm, where a higher score is equal to a higher pain level.
  units on a scale | 63.3 (11.0) | 63.3 (11.3) | 63.8 (11.3) | 63.4 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC Pain Score at 26 Weeks (ITT Population)
Description: The change from baseline in knee pain as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal group to the TH group. The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the change from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat Population - all enrolled subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
units on a scale | -46.4 (19.9) | -46.6 (19.1) | -45.0 (21.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.5874, ANOVA

2. Secondary Outcome: Change From Baseline in WOMAC Pain Score at 3 Weeks (ITT Population)
Description: The change from baseline in knee pain as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal group to the Monovisc group. The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the change from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 3 weeks
Population: Intent to Treat Population (ITT): all enrolled subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
score on a scale | -42.6 (20.0) | -39.5 (20.4) | -41.3 (19.7)
Statistical Analysis 1: Comparison: Cingal vs Monovisc; Test type: Superiority; p = 0.0829, ANOVA

3. Secondary Outcome: OMERACT-OARSI Responder Index at 26 Weeks Post Treatment Comparing the Cingal Group to the TH Group (ITT Population)
Description: The responder rate as identified by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) responder index at 26 weeks post treatment comparing the Cingal® group to the TH group. The OMERACT-OARSI responder index is a proportion of subjects that met the criteria to be a responder.
Time Frame: 26 weeks
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
percentage of subjects | 91.24 | 93.63 | 94.59
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.4673, ANOVA

4. Secondary Outcome: Change From Baseline in WOMAC Physical Function Score at 26 Weeks (ITT Population)
Description: The change from baseline of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Score comparing the Cingal and TH arms (ITT Population). The WOMAC Physical Function Score is a validated visual analog scale from 0 = no limitations in function to 100 mm = highest limitations in function. A negative number for the change from baseline indicates improvement in physical function. A greater negative difference from baseline means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
units on a scale | -42.6 (2.85) | -42.4 (2.85) | -42.4 (2.85)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.9408, ANOVA

5. Secondary Outcome: Change From Baseline in WOMAC Stiffness Score at 26 Weeks (ITT Population)
Description: The change from baseline in knee stiffness as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score comparing the Cingal group to the TH group. The WOMAC Stiffness Score is a validated visual analog scale from 0 = no stiffness to 100 = highest stiffness level. A negative number for the change from baseline indicates reduction in knee stiffness. A greater negative difference from baseline means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
units on a scale | -39.4 (3.17) | -41.1 (3.17) | -38.5 (3.17)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.7770, ANOVA

6. Secondary Outcome: Change From Baseline in Total WOMAC Score at 26 Weeks (ITT Population)
Description: The change from baseline in Total Score as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) comparing the Cingal group to the TH group. The Total WOMAC Score combines the three 0-to-100 point scores from the WOMAC Pain Score, the WOMAC Stiffness Score, and the WOMAC Physical Function Score for a Total Score from 0 = no symptoms to 300 = highest degrees of pain, stiffness, and functional limitation symptoms. A negative number for the change from baseline indicates reduction in pain, stiffness and function limitations. A greater negative difference from baseline means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Triamcinolone Hexacetonide (TH): 20 mg/ml supplied as 1 mL unit dose in a glass ampoule.
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
score on a scale | -128.3 (8.03) | -130.1 (8.03) | -125.9 (8.03)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.7590, ANOVA

7. Secondary Outcome: Change From Baseline in Patient Global Assessment at 26 Weeks (ITT Population)
Description: The change from baseline in the Patient Global Assessment (PGA) between the Cingal and TH arms (ITT population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your index knee bothers you, what is your assessment of how much your knee is bothering you today?" The PGA is scored on a visual analog scale, where 0 = the patient is not bothered to 100 mm = the patient is bothered to the highest degree. A negative number for the change from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat (all enrolled subjects)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
score on a scale | -37.2 (3.37) | -37.3 (3.37) | -37.9 (3.37)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.8309, ANOVA

8. Secondary Outcome: Change From Baseline in the Evaluator Global Assessment at 26 Weeks (ITT Population)
Description: The change from baseline in the Evaluator Global Assessment between the Cingal and TH arms (ITT population). The Evaluator Global Assessment is completed by the Blinded Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the change from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 26 weeks
Population: Intent to Treat (all enrolled subjects)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
score on a scale | -37.4 (2.73) | -36.4 (2.73) | -38.8 (2.73)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.6215, ANOVA

9. Secondary Outcome: Change From Baseline in WOMAC Pain Score at 1 Week (ITT Population)
Description: as for outcome 2
Time Frame: 1 week
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Triamcinolone Hexacetonide: Triamcinolone hexacetonide (TH) is a corticosteroid supplied in a 20 milligram per 1 milliliter (20 mg/mL) intra-articular injection.
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide
Number analyzed (Participants) | 251 | 251 | 74
score on a scale | -35.3 (20.7) | -33.0 (21) | -34.5 (20.7)
Statistical Analysis 1: Comparison: Cingal vs Monovisc; Test type: Superiority; p = 0.2160, ANOVA

10. Secondary Outcome: The Usage of Rescue Medication (Acetaminophen) Through 26 Weeks (ITT Population)
Description: The usage of rescue medication (acetominophen) through 26 weeks post treatment in the Cingal group compared to the TH group using the ITT population.
Time Frame: 26 weeks
Population: Intent to Treat Population (ITT) - all enrolled subjects
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 251 | 251 | 74
pills | 5.4 (19.3) | 5.9 (16.0) | 6.3 (17.0)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.7026, ANOVA

11. Other Pre Specified Outcome: Change From Baseline in WOMAC Pain Score at 3 Weeks in the Per-Protocol Population
Description: as for outcome 2
Time Frame: 3 Weeks
Population: Per-Protocol Population (PP): The PP Population was defined as all subjects who completed the 26 Week Visit (since the primary end point was at 26 Weeks) and have no major protocol violations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 238 | 244 | 69
score on a scale | -43.4 (19.6) | -39.8 (20.4) | -42.5 (18.1)
Statistical Analysis 1: Comparison: Cingal vs Monovisc; Test type: Superiority; p = 0.0438, ANOVA

ADVERSE EVENTS:
Time Frame: All Adverse Events that occurred after signing the Informed Consent Form to 26 weeks post treatment were recorded for all enrolled subjects (Safety Population).
Description: The definitions used for an adverse event and/or serious adverse event are consistent with the definitions used in clinicaltrials.gov.
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/251 | 0/74
Serious Adverse Events (participants affected / at risk) | 7/251 | 0/251 | 0/74
Other Adverse Events (participants affected / at risk) | 101/251 | 101/251 | 20/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=251) | Monovisc (N=251) | Triamcinolone Hexacetonide (TH) (N=74)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Fracture of lateral malleolus, closed (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Delirium tremens (General disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
Varicose Vein (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — The AE is resolved without sequelae
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=251) | Monovisc (N=251) | Triamcinolone Hexacetonide (TH) (N=74)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Palpitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) — Mild
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Glucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Lens dislocation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Mild
Abdominal Pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) — Mild and Moderate
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Diarrhea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) — Mild
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Toothache (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) — Mild
Asthenia (General disorders) | 1 (2) | 0 (0) | 0 (0) — Mild
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Injection site pain (General disorders) | 8 (8) | 7 (8) | 1 (1) — Mild and Moderate
Injection site reaction (General disorders) | 1 (1) | 2 (2) | 0 (0) — Mild
Injection site reaction (General disorders) | 2 (2) | 1 (1) | 0 (0) — Moderate
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Pyrexia (General disorders) | 3 (4) | 0 (0) | 0 (0) — Mild
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Mild
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) — Mild
Bronchitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) — Moderate
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Mild
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Moderate
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Mild
Herpes zoster (General disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Influenza (General disorders) | 2 (2) | 4 (6) | 1 (1) — Mild
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) — Moderate
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) — Mild
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Moderate
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — Mild
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Mild
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 1 (1) — Mild
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — Mild
Viral upper respiratory tract infection (Infections and infestations) | 12 (12) | 16 (18) | 6 (6) — Mild
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Severe
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Mild
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Moderate
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Mild
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Severe
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Mild
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) — Mild
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Moderate
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Mild
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Moderate
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Moderate
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Mild
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — Mild
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) — Mild
Culture urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) — Mild
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (29) | 12 (40) | 2 (2) — Mild
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (19) | 5 (11) | 2 (2) — Moderate
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Severe
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (6) | 1 (1) — Mild
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 0 (0) — Mild
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Joint range of motion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Joint range of motion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Mild
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) — Mild
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) — Moderate
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) — Mild
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 0 (0) — Mild
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 3 (3) — Mild
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 — Moderate
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Severe
Headache (Nervous system disorders) | 31 (47) | 28 (78) | 6 (11) — Mild
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) — Mild
Migraine (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) — Mild
Sciatica (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) — Mild
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Severe
Mental disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Severe
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Benign Prostatic hyperplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Ovulation pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Pneumonitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Moderate
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) — Moderate
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Severe
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Mild
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Moderate
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Moderate
Hypertention (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Mild

LIMITATIONS AND CAVEATS:
Cingal 16-02 did not include a placebo arm, and was an all-active trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03191903/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT03191903/SAP_001.pdf